CLINICAL TRIAL: NCT05000320
Title: VIGAB-BIOSTAT: Neuronal Injury Panel Substudy
Status: Withdrawn | Type: Observational
Why Stopped: study never open to accrual and no subjects were enrolled
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: VIGAB-BIOSTAT; IRB202101781 (Other: UF IRB-01); OCR41006 (Other: UF OnCore)
Record Dates: First submitted 2021-08-10; First posted 2021-08-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2022-09

CONDITIONS: Status Epilepticus; Cardiac Arrest With Successful Resuscitation
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vigabatrin-naive: Adults 18 - 80 years of age suffering from post anoxic status epilepticus (PASE) who have not received vigabatrin.
  Interventions: Diagnostic Test: Neuronal Injury Panel

INTERVENTIONS:
Diagnostic Test: Neuronal Injury Panel — A panel of neuronal and astroglial assays that may be a marker of brain injury.

SUMMARY:
The purpose of this substudy is to collect and analyze control data to characterize the degree of neuronal injury in PASE patients who have not received vigabatrin to later compare with patients who received this therapy and expand data on the utility of the neuronal injury panel for neuroprognostication. Data from this cohort will be compared with the data generated by the treatment cohort in the main VIGAB-STAT study.

DETAILED DESCRIPTION:
Post anoxic status epilepticus (PASE) is the development of intractable seizures in the post-cardiac arrest period once return of spontaneous circulation (ROSC) has been achieved. Historically, this condition has resulted in nearly 100% mortality, and the subset of patients diagnosed with PASE has been excluded from previous therapeutic trials in status epilepticus. The administration of vigabatrin, a GABA-ergic medication that blocks GABA catabolism, is being investigated as an adjunctive therapy to improve neurologic outcomes in this patient population through the VIGAB-STAT program at the University of Florida.

Neuroprognostication in cardiac arrest patients remains imprecise. Outcomes following cardiac arrest depend on a multitude of factors, from details of cardiac arrest (e.g., downtime and rhythm on arrest) to other factors that influence secondary brain injury-all of which are hard to ascertain from objective clinical and laboratory data. Neuronal and astroglial protein assays have been investigated in this patient population as a novel method of quantifying the degree of neuronal injury and may serve as an objective informant of ongoing secondary brain injury, thus being a helpful neuroprognostic tool. This assay can also demonstrate objectively if a neuroprotectant therapy mitigates secondary brain injury and decreases the overall hypoxic-brain injury burden. However, normative data on these assays on post-cardiac arrest patients suffering PASE are lacking.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study, subjects must be 18 - 80 years of age
* Non-traumatic cardiac arrest (regardless of non-perfusing rhythm, etiology, or location of arrest) in whom the decision to treat unequivocal electrographic SE (as defined by the American Clinical Neurophysiology Society: having generalized spike/sharp-wave discharges ≥ 3Hz or any evolving pattern reaching > 4Hz, lasting ≥ 10 minutes, or comprising > 50% of any hour of recording) has been made,
* Requiring anesthetic infusion for any reason,
* Have reliable arterial access for frequent blood sampling
* Be enrolled and have the first specimen drawn within 48 hours of PASE onset.

Exclusion Criteria:

* Subjects must not have a prior history of generalized epilepsy
* Be pregnant or
* Have PASE onset preceding initiation of EEG monitoring.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18-80 years of age suffering from post anoxic status epilepticus (PASE)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-08-17 (Estimated); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
Measure the degree of brain injury | Days 1 - 5
  A neuronal Injury panel of assays will be conducted that may be used to measure the degree of brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Maciel, MD, MSCR, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legriel S, Hilly-Ginoux J, Resche-Rigon M, Merceron S, Pinoteau J, Henry-Lagarrigue M, Bruneel F, Nguyen A, Guezennec P, Troche G, Richard O, Pico F, Bedos JP. Prognostic value of electrographic postanoxic status epilepticus in comatose cardiac-arrest survivors in the therapeutic hypothermia era. Resuscitation. 2013 Mar;84(3):343-50. doi: 10.1016/j.resuscitation.2012.11.001. Epub 2012 Nov 9. PMID 23146879
- [Background] Backman S, Westhall E, Dragancea I, Friberg H, Rundgren M, Ullen S, Cronberg T. Electroencephalographic characteristics of status epilepticus after cardiac arrest. Clin Neurophysiol. 2017 Apr;128(4):681-688. doi: 10.1016/j.clinph.2017.01.002. Epub 2017 Jan 21. PMID 28169132
- [Background] Huesgen KW, Elmelige YO, Yang Z, Chowdhury MAB, Gul S, Maciel CB, Elie-Turenne MC, Becker TK, Cohen SA, Holland A, Montero C, Zhu T, Wang KK, Tyndall JA; Florida Cardiac Arrest Resource Team. Ultra-early serum concentrations of neuronal and astroglial biomarkers predict poor neurological outcome after out-of-hospital cardiac arrest-a pilot neuroprognostic study. Resusc Plus. 2021 Jun 8;7:100133. doi: 10.1016/j.resplu.2021.100133. eCollection 2021 Sep. PMID 34223394
- [Background] Wang KK, Yang Z, Zhu T, Shi Y, Rubenstein R, Tyndall JA, Manley GT. An update on diagnostic and prognostic biomarkers for traumatic brain injury. Expert Rev Mol Diagn. 2018 Feb;18(2):165-180. doi: 10.1080/14737159.2018.1428089. Epub 2018 Jan 23. PMID 29338452